CLINICAL TRIAL: NCT04741854
Title: Development of Advanced Leak Detection Technologies for Positive Airway Pressure Devices Therapies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLP-20-04-01
Record Dates: First submitted 2021-01-11; First posted 2021-02-05 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Investigational Device (Experimental): Participants will be asked to take home the investigational device to use at night while they sleep in place of their own device. The participant's therapy and comfort settings will be copied from their own device to the investigational device.
  Interventions: Device: Positive Airway Pressure (PAP) Therapy

INTERVENTIONS:
Device: Positive Airway Pressure (PAP) Therapy — PAP therapy supplies pressurized air from the flow generator to the upper airway via air tubing and a mask to prevent the repetitive collapse of the upper airway during sleep.

SUMMARY:
This study will take between 1-2 months (with first patient first visit to last patient last visit). Each participant will use the supplied PAP device and mask for a period of up to 14 nights. Participants will complete a series of questionnaires. The study will collect data to support the development of an advance leak detection technology.

DETAILED DESCRIPTION:
The investigation device is designed to collect leak patterns which will be analysed to develop an advanced leak detection technology to help users/patients to troubleshhot therapy issues.

This will be a multi-centre, multiphase, single arm study. The study will be conducted in the home environment.

Recruitment Recruitment will be done via phone calls/ SMS messages/ emails. Participants will be explained the details of the trial and those who wish to take part will be invited to ResMed for the first study visit.

Visit 1 Participants will provide written informed consent. If eligible, baseline participant demographics will be collected. Participants will be shown the investigation equipment. If the participant is happy to proceed, the therapy and comfort settings of the trial PAP device will be set-up to match their current PAP device and a mask similar to the participant's current mask will be provided to take home and be use in place of their own equipment.

Visit 2 After completing 7 days of the trial participants will return to the ResMed. The researcher will review the questionnaire and data quality with the participant.

Visit 2 may not be performed or completed via digital platform. For Phase 2 of this study. Visit 2 may not be completed as confidence in the system set up is achieved via Phase 1.

Visit 3

After completing another 7 days of the trial, participants will return to the ResMed. The participant will return all trial equipment researcher. The participants' questionnaire responses and data will be reviewed. This concludes the participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to give written informed consent.
* Patients who have a possible risk of mouth leak.
* Patients willing to give written consent for the recording of full band audio during sleep session.
* Patients who are willing to not wearing chin strap for a period of nights during study, if they currently use one.
* Patients who can read and comprehend English
* Patients who ≥ 18 years of age
* Patients being established on PAP therapy for the treatment of OSA for ≥ 6 months
* Patients currently using an appropriate mask system, AirFit P10, AirFit N20, AirFit N20, AirFit N30i (2 check version is correct) or similar mask (non-full face).
* Patients who can trial the investigational device for up to 14 nights
* Patients who have been compliant to therapy for the previous 7 nights of use.

Exclusion Criteria:

* Patients willing to give written informed consent.
* Patients who have a possible risk of mouth leak.
* Patients willing to give written consent for the recording of full band audio during sleep session.
* Patients who are willing to not wearing chin strap for a period of nights during study, if they currently use one.
* Patients who can read and comprehend English
* Patients who ≥ 18 years of age
* Patients being established on PAP therapy for the treatment of OSA for ≥ 6 months
* Patients currently using an appropriate mask system, AirFit P10, AirFit N20, AirFit N20, AirFit N30i (2 check version is correct) or similar mask (non-full face).
* Patients who can trial the investigational device for up to 14 nights
* Patients who have been compliant to therapy for the previous 7 nights of use.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Acoustic signals | 2 Months
  Cross-correlation of acoustic signals recorded from the patient environment and the objective leak data recorded by the investigational Positive Airway Pressure Device.

CONTACTS AND LOCATIONS:
Locations (1):
- ResMed BELLA VISTA, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No